CLINICAL TRIAL: NCT03985501
Title: DREPAMASSE Study - Evaluation of a Newborn Screening for Sickle Cell Disease by Tandem Mass Spectrometry
Acronym: DREPAMASSE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0338; 2019-A01346-51 (Other: ID-RCB)
Record Dates: First submitted 2019-06-06; First posted 2019-06-13 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Sickle Cell Disease; Infant, Newborn, Disease; Drepanocytosis
MeSH Terms: conditions — Anemia, Sickle Cell; Disease; Sickle Cell Trait

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- newborn screening for sickle cell disease: Newborns with a targeted neonatal screening for sickle cell disease carried out at the University Hospital of Lyon
  Interventions: Other: SCD newborn screening with the MS/MS method from Zentech

INTERVENTIONS:
Other: SCD newborn screening with the MS/MS method from Zentech — The analysis of the SCD newborn screening with the MS/MS method from Zentech will be realized after achievement and biological validation of the SCD newborn screening in the usual care pathway. The results will be compared with the method used at the Lille Academic Hospital (CHU Lille) (sub-contractor for SCD newborn screening of Lyon)

SUMMARY:
Three methods are actually used in newborn screening for sickle cell disease (SCD) in France: isoelectric focusing, high performance liquid chromatography and capillary electrophoresis. New technologies are currently under development such as Matrix Assisted Laser Desorption Ionisation - Time of Flight (MALDI-TOF) and tandem mass spectrometry (MS/MS) using the SpOtOn Diagnostics Reagent Kit available in United Kingdom only.

Zentech company (Liège, Belgium) is developing a package for SCD newborn screening using MS/MS technology. The main objective of the present study will be to compare this new technique with the technique actually used in the hospital center of Lille (sub-contractor for SCD newborn screening of Lyon) and the haemoglobin analysis to test its accuracy (sensitivity and specificity).

ELIGIBILITY:
Inclusion Criteria:

* Infants with SCD newborn screening conducted in the hospital center of Lyon

Exclusion Criteria:

* Insufficient quantity of sampling
* Parents' opposition to their newborn's participation in the study

Ages: 1 Day to 27 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with SCD newborn screening conducted in the hospital center of Lyon
Sampling Method: Non-Probability Sample
Enrollment: 1431 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Percent agreement between the two techniques | 6 months
  Non-inferiority (difference <1%) in terms of sensitivity and specificity between the results obtained with the MS/MS method and those obtained with the technique currently used at the Lille CHU (sub-contractor for SCD newborn screening of Lyon)

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Groupement Hospitalier Est - Hospices Civils de Lyon, Bron
  - Hopital de la Croix Rousse, Lyon
  - Centre Hospitalier Lyon Sud, Pierre-Bénite